CLINICAL TRIAL: NCT00240357
Title: Open Label Primary Care Study: Rosuvastatin Based Compliance Initiatives Linked To Achievement of LDL Goals. - Denmark
Brief Title: Effect of an Internet Based Compliance Enhancement Tool in Subjects With Hypercholesterolemia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study cancelled prior to FSI
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3560L00002; Orbital
Record Dates: First submitted 2005-10-16; First posted 2005-10-18 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

INTERVENTIONS:
Procedure: Lifestyle Regulation

SUMMARY:
The purpose of the study is to determine whether an Internet based compliance tool is superior to common diet counselling in patients with hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Available personal mailbox and access to the Internet
* Primary hypercholesterolemia with CV risk > 20% over 10 years judged by the investigator or a history of ischemic heart disease or other established atherosclerotic disease (claudicatio intermittens, apoplexia cerebri (ischaemic stroke)) or stable diabetes mellitus
* Fasting LDL-C level > 3.2 mmol/L

Exclusion Criteria:

* Known heterozygous or homozygous familial hypercholesterolemia or known type III hyperlipoproteinaemia (familial dysbetalipoproteinaemia)
* Documented secondary hypercholesterolemia of any cause except stable diabetes mellitus (type 1 or type 2)
* History of serious adverse effect or hypersensitivity reactions to statins, in particular any history of myopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1175
Dates: Start 2003-02

PRIMARY OUTCOMES:
The primary endpoint is the number and percentage of subjects from each group (rosuvastatin or rosuvastatin + a compliance enhancement tool) who reached the DSAM LDL-C target goal (LDL-C < 3.0 mmol/L) after 6 months therapy (24 weeks).

SECONDARY OUTCOMES:
Number and percentage of subjects within the DSAM LDL-C target goal after 3 months therapy
Compliance with study drug assessed by tablet count data
Number and percentage of subjects increasing rosuvastatin dosage from 10 mg to 20 mg at week 12
Percentage change in TC, HDL-C, LDL-C, TG from week 0 to week 24
Change in weight after 6 months therapy
Change in waistline after 6 months therapy

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Denmark Medical Director, MD, Study Director — AstraZeneca A/S
Locations (109):
- Denmark (109):
  - Research Site, Aabenraa
  - Research Site, Aalborg
  - Research Site, Aarhus C
  - Research Site, Aerup
  - Research Site, Albertslund
  - Research Site, Ans
  - Research Site, Ålbæk
  - Research Site, Ålestrup
  - Research Site, Bagsværd
  - Research Site, Billund
  - Research Site, Birkeroed
  - Research Site, Broendby Strand
  - Research Site, Broenshoej
  - Research Site, Copenhagen V
  - Research Site, Elsingore
  - Research Site, Farum
  - Research Site, Fredericia
  - Research Site, Frederiksberg C
  - Research Site, Frederikshavn
  - Research Site, Frederikssund
  - Research Site, Gentofte Municipality
  - Research Site, Glesborg
  - Research Site, Glostrup Municipality
  - Research Site, Goerlev Sjaelland
  - Research Site, Grenå
  - Research Site, Greve
  - Research Site, Grindsted
  - Research Site, Hadsund
  - Research Site, Haslev
  - Research Site, Hårlev
  - Research Site, Hedehusene
  - Research Site, Hellerup
  - Research Site, Helsinge
  - Research Site, Herning
  - Research Site, Hilleroed
  - Research Site, Hoeng
  - Research Site, Hoersholm
  - Research Site, Holbæk
  - Research Site, Hornbæk
  - Research Site, Horsens
  - Research Site, Humlebæk
  - Research Site, Hvidovre
  - Research Site, Ikast
  - Research Site, Jægerspris
  - Research Site, Kalundborg
  - Research Site, Karlslunde
  - Research Site, Kåstrup
  - Research Site, Kjellerup
  - Research Site, Kokkedal
  - Research Site, Kolding
  - Research Site, Kongens Lyngby
  - Research Site, Kværndrup
  - Research Site, Langeskov, Fyn
  - Research Site, Lyngby
  - Research Site, Lystrup
  - Research Site, Maeloev
  - Research Site, Middelfart
  - Research Site, Morud
  - Research Site, Noerre Alslev
  - Research Site, Noerresundby
  - Research Site, Nyborg
  - Research Site, Nykoebing F
  - Research Site, Nærum
  - Research Site, Næstved
  - Research Site, Nørre Broby
  - Research Site, Odense C
  - Research Site, Odense NV
  - Research Site, Oelstykke
  - Research Site, Oksboel
  - Research Site, Randers
  - Research Site, Risskov
  - Research Site, Roedovre
  - Research Site, Roskilde
  - Research Site, Roslev
  - Research Site, Rudkoebing
  - Research Site, Rungsted Kyst
  - Research Site, Sakskoebing
  - Research Site, Saltum
  - Research Site, Skals
  - Research Site, Skive
  - Research Site, Skovlunde
  - Research Site, Slagelse
  - Research Site, Snekkersten
  - Research Site, Soendersoe
  - Research Site, Solroed Strand
  - Research Site, Soroe
  - Research Site, Stege
  - Research Site, Stenlille
  - Research Site, Struer Municipality
  - Research Site, Svendborg
  - Research Site, Svenstrup
  - Research Site, Sæby
  - Research Site, Sønderborg
  - Research Site, Taastrup
  - Research Site, Thorsoe
  - Research Site, Toelloese
  - Research Site, Toender
  - Research Site, Ullerslev
  - Research Site, Vaerloese
  - Research Site, Vanloese
  - Research Site, Varde
  - Research Site, Vedbæk
  - Research Site, Vejle
  - Research Site, Viborg
  - Research Site, Viby J
  - Research Site, Vinderup
  - Research Site, Virum
  - Research Site, Viuf
  - Research Site, Vojens